CLINICAL TRIAL: NCT00970840
Title: Acceptability of Lipid-based Nutrient Supplements (LNS) for Women and Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 200917060-1
Record Dates: First submitted 2009-09-01; First posted 2009-09-03 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2009-09

CONDITIONS: Anemia; Malnutrition
Keywords: Acceptability; Supplements; Home-fortification
MeSH Terms: conditions — Anemia; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LNS-20gM or LNS-P&L (Experimental)
  Interventions: Dietary Supplement: LNS-20gM or LNS-P&L

INTERVENTIONS:
Dietary Supplement: LNS-20gM or LNS-P&L — Participants consumed a test meal (45 g or 50 g) consisting of LNS-20gM or LNS-P&L mixed with fermented maize porridge, after which they were provided with the respective LNS supplements for use at home daily for 14 d

SUMMARY:
Inadequate micronutrient intakes during pregnancy, lactation and infancy remain a major problem in Ghana. Lipid-based nutrient supplements (LNS) made using vegetable oil, groundnut paste, milk, sugar, and micronutrients may offer a solution.

The proposed study will test the acceptability of a lipid-based nutrient supplement designed for infants (LNS-20gM) and another designed for pregnant and lactating women (LNS-P&L). Participants will consume a test meal consisting of LNS-20gM (20 infants) or LNS-P&L (20 pregnant and lactating women) mixed with fermented maize porridge, after which they will be given the respective LNS supplement for use at home for 14 d. Primary outcome is the proportion of the test-meal consumed. The investigators hypothesize that subjects will consume at 75% of the test meal offered.

DETAILED DESCRIPTION:
This study is a taste test to confirm the acceptability of lipid-based nutrient supplements (LNS), which are semi-solid pastes comprising groundnut paste, milk, sugar, vegetable oil and micronutrients, for home fortification of foods consumed by infants and by pregnant and lactating women. Two types of supplements will be evaluated, one for infants (LNS20gM) and one for pregnant and lactating women (LNS P&L). The LNS-20gM is similar to the Nutributter we used previously in Ghana and provides generally the Recommended Nutrient Intakes (RNI) for 18 vitamins and minerals for infants from 6 to 18 mo of age. The LNS-P&L is modeled on the UNICEF/WHO/UNU international multiple micronutrient preparation (UNIMMAP) for pregnant and lactating women and similar products used in Guinea Bissau. Each supplement (20 g/day) will provide 118 kcal/day.

Procedures:The study will be carried out in two phases. The first test trial will be conducted within the premises of the Maternal and Child Health Clinics, where study participants will be recruited.

Potential study participants or their mothers (in the case of infants) will be asked verbally using a screening questionnaire at the time of recruitment if they are known to be intolerant to peanut or milk products, in which case they will be excluded. Because infants must have been receiving complementary foods at least 30 days prior to taking part in the study, this will not be too difficult to find out. For subjects unaware of whether they are intolerant to peanut or milk products, they will be asked not to go home immediately after finishing the experiment, but to continue to remain in (or around) the testing room for at least one hour whilst the study staff keep watch. Should there be any skin, respiratory or gastrointestinal symptoms in any subject during that time, they will be immediately referred to the hospital. When leaving the testing room for the home, those subjects (or their mothers) will be given the project's mobile phone number to call in case there are any symptoms during the next few hours.

Potential subjects or their mothers (in the case of infants) will be asked if they feel ill using the screening questionnaire. Subjects who report any feeling of illness will be excluded. The Maternal and Child Health clinics (MCH) where subjects will be recruited provide mainly routine services for women (such as ante-natal services for pregnant women) and children (such as weight monitoring and promotion and vaccination). We expect that nearly all women and infants attending these clinics will be apparently in good health and not ill.

Phase 1 - Test-feeding:

Study participants will be women (n = 20) ≥ 18 y of age who are either pregnant (n = 10) or lactating (n = 10) and infants (n = 20 accompanied by their mothers) 6 - 12 mo of age randomly-selected from Maternal and Child Health clinics in Manya and Yiko Krobo districts of the Eastern Region of Ghana. All subjects must be apparently healthy and must not have eaten any food (including breast milk) during the previous one hour.

1. Test-feeding of LNS P&L:

   After consent, pregnant (n=10) and lactating women (n=10) will be asked to come to the clinic the next day for an orientation session during which background data will be collected and the experimental procedures will be practiced including tasting of the food and completion of the tasting questionnaire. The second day will be Test Day 1, during which the actual tasting will be recorded. Women will be asked to consume 45 g of koko mixed with LNS P&L (prepared from mixing 150 g LNS-P&L with 600 g fresh koko with moisture content of about 90%). Time taken to consume the entire amount, or proportion of the amount consumed within 15 minutes, will be measured. Women will be asked to rate the mixture's appearance, aroma, flavor, consistency and overall degree of liking using a hedonic scale. On the third day (Test Day 2) of the trial, the above procedures will be repeated using koko mixed with Nutributter instead.

   Koko for the test feeding will be provided by the project. Project staff will purchase fermented dough (the main ingredient) from the local market to prepare the koko under good hygienic conditions in our project house. After preparation, the koko will be kept hot in a thermos flask prior to being served to study participants at the MCH clinic. Between the time the koko is prepared and the time the test feeding is completed, which will take 2-3 hours, the koko can be kept at a temperature of 70 - 90 °C inside the thermos flask to prevent bacterial contamination. The Nutributter and the LNS supplements will be commercially produced by Nutriset SAS (Malaunay, France) and provided to the Project for testing.
2. Test-feeding of LNS20gM:

After consent, the mother (or care-taker) of each participating infant will be asked to come to the clinic with the child the next day for an orientation session during which background data will be collected and the experimental procedures will be practiced including tasting of the food and completion of the tasting questionnaire. The second day will be Test Day 1, during which the actual tasting will be recorded. Mothers or caretakers will be given 50 g of koko mixed with LNS 20gM (prepared from mixing 150 g LNS-20gM with 600 g fresh koko with moisture content of about 90%). They will be asked to consume one teaspoon of the mixture (~ 5 g), and then feed the rest (~ 45 g) to their infants after it is re-weighed. During this time, the child should be awake and alert, and either calm or fussy - but not drowsy or crying. Time taken by the child to consume the remaining portion, or proportion consumed by the child within 15 minutes, will be measured. The mother or caretaker will then rate the mixture's appearance, aroma, flavor and consistency based on her own opinion, and her perception of the infant's degree of liking. Mothers will be asked to report to us if the child vomits in the next hour, or develops any new symptoms such as rash or wheezing. On the third day (Test Day 2) of the trial, the above procedures will be repeated using koko mixed with Nutributter instead.

Phase 2 - Assessment under real-life conditions:

Pregnant and lactating women who participated in the Phase 1 trial will be given a two-week supply of LNS P&L, which they will add to their prepared food daily during the two-week period. Mothers of children who participated in the Phase 1 trial will receive LNS20gM, which they will add to their infants' prepared food for 2 weeks. The dose for LNS P&L or LNS20gM is 20 g/day. To ensure that subjects consume the entire daily dose, women will be instructed, as done previously in our study in Ghana, to mix their own or their infant's daily dose with 2-3 tablespoons of the food, to be consumed before consuming the rest of the food.

Dosage and directions for use will be as follows: 20 g (~4 teaspoons) per day divided into 2 portions and consumed at two different times of the day (2 x 2 teaspoons). Mix the portion of the supplement to be consumed with 2-3 tablespoons of the already prepared food, and eat the mixture before eating the rest of the food. Do not cook food with the supplement. Store supplement at room temperature. There is no need for refrigeration.

A structured questionnaire will be used to gather background information on socioeconomic status, and maternal and infant feeding behavior. The amount of LNS consumed by subjects will be monitored weekly, and the reactions to the products will be obtained at the end.

ELIGIBILITY:
Inclusion Criteria (infants):

* 6-12 months of age
* currently receiving breast milk
* has been consuming complementary foods for at least 30 days

Inclusion Criteria (women):

* being ≥ 18 years of age
* confirmed to be pregnant or breastfeeding

Exclusion Criteria:

* intolerance to milk or peanut
* illness requiring referral

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2009-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Proportion of test-meal consumed | One day

SECONDARY OUTCOMES:
Degree of liking for appearance, aroma, flavor and consistency of LNS product mixed with koko | 14 days
Amount of LNS consumed during the 14-day study period | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn G. Dewey, PhD, Study Director — UC Davis; Anna Lartey, PhD, Principal Investigator — University of Ghana
Locations (1):
- St. Martins de Porres Hospital, Agomanya, Ghana